CLINICAL TRIAL: NCT03911362
Title: A Comparison of the Effect on Stress Urinary Incontinence of Lumbopelvic Stabilisation Exercises and Pelvic Floor Exercises: A Randomised Controlled Trial
Brief Title: A Comparison of Lumbopelvic Stabilisation and Pelvic Floor Exercises on the Stress Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Meryem Kurek eken, Associated Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/1507
Record Dates: First submitted 2019-03-10; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Stress Urinary Incontinence; Pelvic Floor Disorders
Keywords: Lumbopelvic Stabilisation Exercises; Pelvic Floor Exercises; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbopelvic Stabilisation Exercises (Active Comparator): Starting with co-contraction of the transversus abdominis (TA) muscle and other muscles together with diaphragm breathing, and continuing the exercises with upper and lower extremity movements together with TA and multifidus contraction
  Interventions: Behavioral: Lumbopelvic Stabilisation Exercises Group
- Pelvic Floor Exercises (Active Comparator): The pelvic flor exercise will be in the form of contraction-release for rapidly contracting muscle fibres and for slowly contracting muscle fibres,slow contraction by counting to ten hold for a count of ten, then gradually relax by counting to ten.
  Interventions: Behavioral: Pelvic Floor Exercises Group

INTERVENTIONS:
Behavioral: Lumbopelvic Stabilisation Exercises Group — Lumbopelvic stabilisation exercises will be taught the basic movement, starting with co-contraction of the transversus abdominis (TA) muscle and other muscles together with diaphragm breathing, and continuing the exercises with upper and lower extremity movements together with TA and multifidus contraction.
  Arms: Lumbopelvic Stabilisation Exercises
Behavioral: Pelvic Floor Exercises Group — The pelvic flor exercise will be in the form of contraction-release for rapidly contracting muscle fibres, and for slowly contracting muscle fibres, slow contraction by counting to ten, hold for a count of ten, then gradually relax by counting to ten
  Arms: Pelvic Floor Exercises

SUMMARY:
The patients diagnosed with stress urinary incontinence and included in the study. According to randomisation plan one group will be instructed by a physiotherapist to perform pelvic flor exercises and the other group will be instructed by the same physiotherapist to perform dynamic lumbopelvic stabilisation exercises.Throughout the study, the women will be followed up to ensure the exercises are performed. The exercises will be applied for approximately 30 mins once a day for a period of 10 weeks.

DETAILED DESCRIPTION:
The females included in the study will be separated into 2 groups in the randomisation plan. One group will be instructed by a physiotherapist to perform pelvic flor exercises, and the other group will be instructed by the same physiotherapist to perform dynamic lumbopelvic stabilisation exercises. After a demonstration by the physiotherapist of how both exercises should be performed, the women will be requested to perform the exercises under the supervision of the physiotherapist. The pelvic flor exercise will be in the form of contraction-release for rapidly contracting muscle fibres, and for slowly contracting muscle fibres, slow contraction by counting to ten, hold for a count of ten, then gradually relax by counting to ten. The exercises will start as 5 sets of 10 repetitions per day, then each week the number of sets will be increased by 5 to reach 30 sets per day, and the exercises will be continued at this rate of 30 sets per day.

The women who will perform the dynamic lumbopelvic stabilisation exercises will be taught the basic movement, starting with co-contraction of the transversus abdominis (TA) muscle and other muscles together with diaphragm breathing, and continuing the exercises with upper and lower extremity movements together with TA and multifidus contraction. Initially the exercise position is held for 5-10 secs with 10 repetitions, and as the program advances the time of holding the position will be extended to 30-45 secs. Throughout the study, the women will be followed up to ensure the exercises are performed. The exercises will be applied for approximately 30 mins once a day for a period of 10 weeks.

The Q-Tip test will be used in the evaluation of uretero vesical junction (UVJ) mobility. A cotton swab lubricated with lidocaine gel will be used in the test. The cotton swab will be placed from the external urethral meatus and will be slowly pushed towards the bladder until resistance is felt. This point where resistance is met will be accepted as the UVJ. During the test, the angle will be measured during maximal strain by drawing the labia to the sides.

The patients diagnosed with stress urinary incontinence and included in the study will be taught the lumbopelvic stabilisation and pelvic floor exercises in the clinic under the guidance of the physiotherapist.

Study procedure:

In literature, the physiological effects of the exercises have been reported to emerge 2 weeks after starting and complaints reduce in 6-8 weeks. Therefore the patients will be instructed to perform the lumbopelvic stabilisation exercises at home, once a day for approximately 30 mins for a period of 10 weeks. Similarly the pelvic flor exercises will be performed for 10 weeks, once a day lasting approximately 30 mins. On 2 days a week, the women in both groups will perform the exercises under the guidance of the physiotherapist in the clinic. In this way, the necessary follow-up will be applied that the women are performing the pelvic flor muscle exercises and the lumbopelvic stabilisation exercises correctly and completely.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 35 years
* BMI <29 kg/m2
* Are willing to participate in the research
* Premenopausal
* Able to self-report urine loss
* Educational level of at least primary school
* Positive cough provocation test (stress test)
* Positive Q-tip test,
* No complaints of constipation

Exclusion Criteria:

* Musculoskeletal system disorder
* Neurological dysfunction
* Genital prolapse more then second stage
* Hormone replacement therapy use
* Postmenopausal
* Anticholinergic drug use
* Urge and mixed incontinence
* Diuretic drug use
* Antidepressant drugs use
* Caffeine intake of >4 cups/day
* Diabetes insipidus
* Urinary infection
* Vaginal infection
* History of urinary or genital surgery
* Malignancy
* Pelvic Floor Trauma
* Lumbar disc hernia
* Pregnancy
* Breast-feeding
* Diabetes mellitus
* Hypertension
* BMI>30 kg/m2
* Chronic obstructive sleep apnea
* Chronic lung disease

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 2 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
The primer outcome of the study was to investigate the effects of lumbopelvic stabilisation exercises and pelvic floor exercises on the severity of incontinence in women with a diagnosis of stress urinary incontinence | six month
  The severity of incontinence at before and after the exercises (total exercise duration is 10 weeks) will measure with Urogenital Distress Inventory. The change from baseline in Urogenital Distress Inventory after the exercises intervention will be measured by decrease on the severity of incontinence.
The other primer outcome of the study was to lumbopelvic stabilisation exercises and pelvic floor exercises on the severity of incontinence in women with a diagnosis of stress urinary incontinence | six month
  The severity of incontinence at before and after the exercises (total exercise duration is 10 weeks) will measure with Incontinence Impact Questionnaire. The change from baseline in Incontinence Impact Questionnaire after the exercises intervention will be measured by decrease on the severity of incontinence.
The another primer outcome of the study was to investigate the effects of lumbopelvic stabilisation exercises and pelvic floor exercises on the amount of urinary output in women with a diagnosis of stress urinary incontinence | six month
  The amount of urinary output and urine leakage in women during five days before exercises and five days after exercises (total exercise duration is 10 weeks) will Bladder Diary with measure. The amount of urinary output and urine leakage before and after exercises will be measured by decrease in urination of frequency and urine leakage at Bladder Diary.

SECONDARY OUTCOMES:
The seconder outcome of the study was to investigate the effects of lumbopelvic stabilisation exercise and pelvic floor exercise on the degree of quality of life in women with a diagnosis of stress urinary incontinence | six month
  Quality of life of women will measure with Incontinence Quality of Life Questionnaire. The degree of quality of life will be measured by change from baseline in Incontinence Quality of Life Questionnaire after the exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Kürek Eken, Associate, Study Director — Adnan Menderes University Obstetric Clinic
Locations (1):
- Meryem Kurek EKEN, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322